CLINICAL TRIAL: NCT03574324
Title: A Multicenter, Randomized Controlled Phase III Clinical Trial of TPF Induction Chemotherapy Versus PF Adjuvant Chemotherapy Combined With Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Nasopharyngeal Carcinoma
Brief Title: TPF Induction Chemotherapy vs PF Adjuvant Chemotherapy Combined With Concurrent Chemoradiotherapy in the Treatment of Locally Advanced NPC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Feng Jing, Head and neck cancer director, chief researcher, clinical professor, Guiyang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180602
Record Dates: First submitted 2018-06-02; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPF+CCRT (Experimental): TPF neoadjuvant chemotherapy followed by cisplatin chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Drug: TPF+CCRT
- CCRE+PF (Other): Cisplatin chemotherapy concurrent combined with intensity-modulated radiation therapy followed by PF adjuvant chemotherapy
  Interventions: Drug: CCRT+PF

INTERVENTIONS:
Drug: TPF+CCRT — Patients receive Neoadjuvant Docetaxel (75mg/m2 on day1 03:30-04:30) and cisplatin (75mg/m2 on day 1-5 10:00-22:00) and 5-FU(750mg/m2 on day 1-5 22:00-10:00) every 21days for three cycles followed by concurrent cisplatin (100mg/m2 on day1 10:00-22:00)every 21 days for three cycles during radiotherapy
  Other Names: Experimental group
  Arms: TPF+CCRT
Drug: CCRT+PF — Patients receive concurrent cisplatin (100mg/m2 on day1 10:00-22:00)every 21 days for three cycles during radiotherapy followed by adjuvant cisplatin (80mg/m2 on day 1-5 10:00-22:00) and 5-FU(800mg/m2 on day 1-5 22:00-10:00) every 21days for three cycles
  Other Names: Control group
  Arms: CCRE+PF

SUMMARY:
Through randomized controlled phase III multicenter clinical trials, TPF induction chemotherapy vs. PF regimen adjuvant chemotherapy concurrently Radiotherapy and chemotherapy for the treatment of locally advanced nasopharyngeal carcinoma: the efficacy, toxicity and quality of life, and further improvement Survival rate and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).
2. Clinical staged as III，IVa（according to the American Joint Committee on Cancer(AJCC) 7th edition）
3. Fertility women should ensure contraception during entry into the study.
4. Age 18-69 years old.
5. Karnofsky scale(KPS)≥70.
6. Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
7. Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
8. Adequate renal function: creatinine clearance ≥60 ml/min.
9. Patients must be informed of the investigational nature of this study and give written informed consent

Exclusion Criteria:

1. With distant metastasis.
2. who had received prior chemotherapy or radiotherapy.
3. patients have physical or mental illness, and by researchers believe that patients 4.can not be completely or fully understood in this study possible complications.

5.pregnancy (via the urine or serum β-HCG test confirmed) or during lactation. 6.serious complications, such as uncontrolled hypertension, heart failure, diabetes and so on.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2023-05-24 (Estimated); Study Completion 2023-05-24 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 3 years
  Progress-free survival(year) is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  The OS(year) was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional failure-free survival(LRFS) | 3 years
  The LRFS(year) is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant metastasis-free survival(DMFS) | 3 years
  The DMFS(year) is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Overall response rate | 12 weeks after completion of concurrent chemoradiotherapy
  Tumour response(CR/PR/SD/PD) was classified according to RECIST v1.1
Incidence of acute and late toxicity | 3 years
  Incidence of acute toxicity（Grade1/2/3/4） is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Li, Master, Principal Investigator — Guizhou Provincial Cancer Hospital
Locations (1):
- Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No